CLINICAL TRIAL: NCT04985097
Title: Preliminary Evaluation of the Clinical Benefit of a Novel Visual Rehabilitation System in Patients Implanted With Trifocal Diffractive Intraocular Lenses: A Blinded Randomized Placebo-controlled Clinical Trial
Brief Title: Home-based Visual Training in Patients Implanted With Trifocal Diffractive Intraocular Lenses
Acronym: OPTicTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Increase-Tech (Other)
Collaborators: University of Alicante (Other); Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other); Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASVENM-20-437
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Visual Disturbances and Blindness; Visual Acuity Reduced Transiently
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Intervention Model Description: Experimental group vs control group
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Half an hour of active visual training per day for a period of 20 consecutive days with the Optictrain software
  Interventions: Procedure: Implantation of trifocal diffractive intraocular lenses
- Control group (Sham Comparator): Half an hour of using a videogame without specific stimuli to improve visual performance (Fun Kid Racing 3.53 for Android) per day for a period of 20 consecutive days
  Interventions: Procedure: Implantation of trifocal diffractive intraocular lenses

INTERVENTIONS:
Procedure: Implantation of trifocal diffractive intraocular lenses — Postsurgical monocular and binocular assessment of corrected and uncorrected near, intermediate and distance visual acuity and near and distance mesopic contrast sensitivity before and after the assigned vision training

SUMMARY:
This multicentre randomised controlled trial aimed to reduce the visual discomfort that patients implanted with trifocal diffractive intraocular lenses may experience after surgery. To this end, a visual training software (Optictrain) was developed in which Gabor patches were presented to the patient on a hand-held electronic device. Patients who met all inclusion criteria and consented to participate underwent half an hour of visual training per day for a period of 20 consecutive days remotely on a colourimetrically characterised Samsung Galaxy Tab A device on which the Optictrain software (n=30) or a placebo software (n=30), respectively, was pre-installed. Corrected and uncorrected near, intermediate and distance visual acuity (VA) and mesopic near and distance contrast sensitivity (CS) were measured monocularly and binocularly at two visits: during the first postoperative week (V0) and after 20 days of visual training with the assigned software (V1). The statistical analysis of the results obtained in the study has not yet been carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 an 90 years
* Patients implanted with trifocal diffractive intraocular lenses
* Availability and motivation to perform the visual training assigned

Exclusion Criteria:

* Age under 18 or over 90 years
* Presence of irregular cornea, illiteracy or cognitive impairment
* History of eye surgery or presence of any active ocular disease
* Intraoperative complications leading to significant visual sequelae
* Patients implanted with monofocal, extended depth of focus or refractive multifocal IOLs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Visual acuity | During the first post-operative week and after 20 days of vision training with the randomly assigned software
  Monocular and binocular corrected and uncorrected visual acuity under near, intermediate and distance conditions
Contrast sensitivity | During the first post-operative week and after 20 days of vision training with the randomly assigned software
  Monocular and binocular mesopic contrast sensitivity under near and distance conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pinero DP, Maldonado-Lopez MJ, Molina-Martin A, Garcia-Sanchez N, Ramon ML, Rincon JL, Holgueras A, Arenillas JF, Planchuelo-Gomez A, Leal-Vega L, Coco-Martin MB. Randomised placebo-controlled clinical trial evaluating the impact of a new visual rehabilitation program on neuroadaptation in patients implanted with trifocal intraocular lenses. Int Ophthalmol. 2023 Nov;43(11):4035-4053. doi: 10.1007/s10792-023-02809-9. Epub 2023 Jul 18. PMID 37464228